CLINICAL TRIAL: NCT04242459
Title: Optimising Radiation Therapy in Head and Neck Cancers Using Functional Image-Guided Radiotherapy and Novel Biomarkers
Acronym: INSIGHT-2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR4934
Record Dates: First submitted 2019-11-08; First posted 2020-01-27 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Cancer
Keywords: Cancer; Oropharynx; HPV; Base of Skull
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will commence with a Feasibility Radiotherapy planning CT study consisting of 13 participants, then will recruit to the the main phase I/II interventional study consisting of 3 independent cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Feasibility Study (No Intervention): This is a radiotherapy planning study to evaluate the feasibility to acquire longitudinal MRI scans during radiotherapy (prior to the main study) thus, participants will receive standard-of-care chemoradiation therapy (CRT) as per departmental protocol without any treatment adaptation.
- HPV associated OPC Participants (Experimental): Participants will be treated initially with the standard radiotherapy dose of:
  * 65 grays (Gy) in 30 fractions (2.17Gy per fraction) over 6 weeks to the primary and nodal tumour.
  * 54Gy in 30 fractions (1.8Gy per fraction) over 6 weeks to the nodal areas at risk of harbouring microscopic disease
  In the 2nd week and 4th week of treatment, the participants will undergo Adaptive Radiotherapy to account for anatomical changes.
  Interventions: Radiation: Adaptive Radiotherapy
- HPV negative OPC Participants - Radiotherapy dose escalation (Experimental): Participants will be treated initially with the standard radiotherapy dose of:
  * 65Gy in 30 fractions (2.17Gy per fraction) over 6 weeks to the primary and nodal tumour.
  * 54Gy in 30 fractions (1.8Gy per fraction) over 6 weeks to the nodal areas at risk of harbouring microscopic disease
  After 10 fractions the participants will be stratified into either "responders" or "non-responders" categories based on Apparent Diffusion Coefficients (ADC) response at week 2 of CRT.
  Participants classified as "responders" will complete treatment without any radiotherapy dose changes. Their radiotherapy treatment target volumes will be adapted at weeks 2 and 4 of CRT to account for volume changes to the tumour.
  The "non-responders" will undergo an increase in dose per fraction to Clinical Target Volume-1 (CTV-1) primary for fractions 11 to 30.
  Interventions: Radiation: Adaptive Radiotherapy
- Base of Skull HNC Participants (Experimental): Participants will be treated initially with the standard radiotherapy dose of:
  * 65Gy in 30 fractions (2.17Gy per fraction) over 6 weeks to the primary and nodal tumour.
  * 54Gy in 30 fractions (1.8Gy per fraction) over 6 weeks to the nodal areas at risk of harbouring microscopic disease
  Participants will undergo standard treatment with 3 cycles of induction chemotherapy followed by chemo-radiotherapy dose. Their radiotherapy treatment will be adapted at weeks 2 and 4 of CRT to account for volume changes to the tumour.
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — Determining the radiotherapy dose delivered to organs at risk (OAR) or to the target volume (dependent on what arm the participant is assigned to) through adaptive radiotherapy volume adaption planning
  Arms: Base of Skull HNC Participants; HPV associated OPC Participants; HPV negative OPC Participants - Radiotherapy dose escalation

SUMMARY:
This is a non-randomised study to develop personalised treatment approaches in participants with Locally Advanced Head and Neck Cancer (HNC) of the oropharynx and base of skull by integrating the use of MR-guided Adaptive Radiotherapy (MRgRT) and functional image-guided radiotherapy (FIgRT).

The study is made up of two parts:

1. Feasibility planning study consisting of a total of 13 patients. This will include patients with either Human papilomavirus-associated (HPV-associated) oropharyngeal cancer (OPC), Human papilomavirus-negative (HPV-negative) OPC or Base of Skull HNC.
2. Single centre prospective interventional phase I/II study (main study) made up of 3 independent arms (on the condition of success of the feasibility stage).

   1. Cohort 1: HPV-associated OPC consisting of 25 participants
   2. Cohort 2: HPV-negative OPC consisting of a minimum of 10 patients and a maximum of 53 participants
   3. Cohort 3: Base of Skull HNC consisting of 25 participants

DETAILED DESCRIPTION:
This study is looking at improving radiotherapy treatment for head and neck cancers by:

1. Repeating the radiotherapy planning scan at weeks 2 and 4 of treatment so that investigators can adapt the radiotherapy to changes to the shape of the cancer and the patient's body. These changes can affect the accuracy and the radiotherapy doses delivered.
2. Using a MR (magnetic resonance) scans to view and target the cancer with more precision.
3. Identifying HPV negative oropharyngeal cancer who are non-responders and increasing the radiotherapy dose.

The 3 groups of patients are:

1. Cancers of the oropharynx (middle of the throat) that test positive for HPV (human papilloma virus). If HPV is present, the cancer responds better to treatment and there is a higher chance of cure. In this group, the investigators aim is to reduce radiotherapy associated long-term side effects by sparing healthy tissue from high doses.
2. If the oropharyngeal cancers test negative for HPV, they are less likely to respond well to treatment. The investigator's department has shown that investigators can predict which patients will respond to treatment using a special type of MR scan. Investigators will increase the dose of radiotherapy to HPV negative patients who are predicted to be non-responders with the aim of improving the chance of cure.
3. Cancers that located at the base of the skull are not seen very well on CT scan. By using MR imaging, investigators can visualize the surrounding normal organs and the cancer better, target the cancer with more precision and adapt to changes to the healthy organs and tumour.

Investigators will also test if they can predict response to treatment by checking blood for fragments of the cancer and using a special MRI.

The study will be conducted at the Royal Marsden in Sutton only and will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Feasibility study and Main Study:

* Participants with stage III/IV ((American Joint Committee (AJC) Tumour, Nodes, Metastasis (TMN) on Cancer Version 7)) head and neck cancer planned for primary radical chemo-radiotherapy OR induction chemotherapy followed by chemoradiotherapy with concomitant platinum-based chemotherapy.
* Age between 18 and 70 years.
* Participant can provide informed consent.
* World Health Organisation (WHO) performance status 0 - 1.
* Creatinine Clearance >50ml/minute
* Absolute Neutrophil Count ≥1.5 x10^9/L
* Platelets ≥100 x10^9/L
* Haemoglobin ≥90g/L

Feasibility Study:

- Participants with either HPV associated OPC, HPV negative OPC or Base of Skull HNC.

Low Risk HPV associated OPC:

* T1-3, N0-2c (AJCC 7th Edition, stage III and above)
* Participants with histologically proven squamous cell carcinoma of the head and neck
* p16 positive (defined as >70% cells staining positive)
* <10 year pack smoking history

HPV Associated OPC:

* Patients with histologically proven squamous cell carcinoma of the head and neck
* T1-3,N0-2c (AJCC 7th Edition, stage III and above) with ≥10 pack/ year smoking history
* p16 positive
* Any T4 and/or N3 regardless of smoking history
* Primary tumour size </=5cm

HPV negative OPC, hypopharyngeal or laryngeal cancer:

* Patients with histologically proven squamous cell carcinoma of the head and neck
* T1-4,N0-3 (AJCC 7th edition, stage III and above)
* p16 negative (if OPC)
* Primary tumour size </=5cm

Base of skull Head and Neck Cancer:

- Participants with histologically proven squamous cell carcinoma or undifferentiated carcinoma of the head and neck (sinonasal and nasopharynx)

Exclusion Criteria:

* WHO performance status >=2.
* Participants with any previous malignancy except non-melanoma skin cancer.
* Participants with prior radiotherapy to the head and neck region
* Participants with contraindications to MRI scan.
* Participants with contraindications to IV contrast agents.
* Participants with renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of participants undergoing MR scan at baseline, week 2 and week 4 and feasibility of producing an adaptive radiotherapy plan | Through feasibility study completion, estimated 6 months.
  To calculate the proportion of participants who have successfully undergone the planned MRI scan at baseline and weeks 2 and 4 to determine the feasibility of producing an adaptive radiotherapy plan in the feasibility study.
Compare the mean cumulative radiotherapy doses Main Study, Cohort 1: Compare the mean cumulative radiotherapy doses received by the parotid gland in an adaptive plan at weeks 3 and 5 to a non-adaptive plan | Through main study treatment period, estimated 5 years.
  To determine the radiotherapy dose delivered to the parotid gland through adaptive radiotherapy volume adaptation planning compared to a non-adaptive radiotherapy approach in the main study, cohort 1.
Assess the safety of radiotherapy dose escalation by measuring the grades of acute radiation induced toxicities using NCI CTCAE v5.0 scores at 3 months | Through main study treatment period, estimated 5 years.
  To assess the safety of radiotherapy dose escalation by measuring the grades of acute radiation induced toxicities which will be assessed using the NCI CTCAE v5.0 scores at 3 months in the main study, cohort 2.
Determine the Maximum Tolerated Dose (MTD) of the escalated radiotherapy dose as per the dose escalation criteria and stopping rules set out in the protocol | Through main study treatment period, estimated 5 years.
  To determine the MTD of the escalated radiotherapy dose in the main study as per the dose escalation criteria and stopping rules as outlined in the protocol in the main study, cohort 2.
Compare the radiotherapy doses to the parotid glands calculated and recorded at baseline with doses from the adaptive plan at weeks 3 and 5 | Through main study treatment period, estimated 5 years.
  To calculate and record radiotherapy doses to the parotid glands at baseline and compare these to doses from the adaptive plan at weeks 3 and 5 in the main study, cohort 3.

SECONDARY OUTCOMES:
Calculate the proportion of patients who investigators can successfully produce an adaptive radiotherapy plan at weeks 3 and 5 within 1 week of their rescan to account for anatomical changes. | Through feasibility study completion, estimated 6 months.
  To calculate the proportion of patients who investigators can successfully produce an adaptive radiotherapy plan at weeks 3 and 5 within 1 week of their rescan to account for anatomical changes.
  To calculate whether investigators can create an adaptive radiotherapy plan at weeks 3 and 5.
Calculate participants complete response rate at 3 months which is defined as no clinically visible, palpable or measurable disease on imaging or no residual tumour on neck dissection or directed biopsy | Through main study treatment period, estimated 5 years.
  To calculate the complete response rate of participants at 3 months in the main study, cohorts 1-3. Response rate is defined as no clinically visible, palpable or measurable disease on imaging (PET-CT and/or MRI) or no residual tumour on neck dissection or directed biopsy.
Calculate the progression free survival which is defined as the time from entry into the study until disease progression or death (days) | Through main study treatment period, estimated 5 years.
  To calculate the progression free survival which is defined as the time from entry into the study until disease progression or death in the main study, cohorts 1-3. This will be measured in whole days.
Calculate the disease specific survival which is defined as the time from entry into the study until death from any cause (days) | Through main study treatment period, estimated 5 years.
  Calculate the disease specific survival which is defined as the time from entry into the study until death from any cause in the main study, cohorts 1-3. This will be measured in whole days.
Assess quality of life using the EORTC Quality of Life Questionnaire (QLQ) C30 version 3.0 with the associated Head and Neck module (HN35) | Through main study treatment period, estimated 5 years.
  Assess quality of life using the EORTC Quality of Life Questionnaire (QLQ) C30 version 3.0 with the associated Head and Neck module (HN35) in the main study, cohorts 1-3.
Assess late radiation induced toxicities which will be recorded using the late effects in normal tissues subjective, objective, management and analytic scales (LENT SOMA) score and NCI CTCAE v5.0 late radiotherapy scoring systems. | Through main study treatment period, estimated 5 years.
  To assess late radiation induced toxicities which will be recorded using the LENT SOMA score and NCI CTCAE v5.0 late radiotherapy scoring systems. The incidence and prevalence (highest grades) of late side effects of radiotherapy will be reported in the main study, cohorts 1-3.
Calculate the duration of acute radiation induced toxicities will be assessed using the NCI CTCAE v5.0 score (HPV associated OPC and skull base tumours); All participants will be evaluated assess xerostomia, mucositis, dysphagia and dermatitis | Through main study treatment period, estimated 5 years.
  To calculate the duration of acute radiation induced toxicities will be assessed using the NCI CTCAE v5.0 score (HPV associated OPC and skull base tumours); All participants will be evaluated using the NCI CTCAE v5.0 score to assess xerostomia, mucositis, dysphagia and dermatitis in the main study, cohorts 1-3.
Assess the Incidence of feeding tube dependency at one year (HPV negative) which is defined as participant needing supplementation of nutrition by feeding tube. | Through main study treatment period, estimated 5 years.
  To assess the Incidence of feeding tube dependency at one year (HPV negative) which is defined as participant needing supplementation of nutrition by feeding tube In the main study, cohorts 1-3.
Calculate the mean radiotherapy doses to the organs at risk (spinal cord, optic chiasm and brainstem) and target volume will be calculated and recorded at baseline and compared to doses from the adaptive plan at weeks 3 and 5. | Through main study treatment period, estimated 5 years.
  To calculate the mean radiotherapy doses to the organs at risk (spinal cord, optic chiasm and brainstem) and target volume will be calculated and recorded at baseline and compared to doses from the adaptive plan at weeks 3 and 5 in the main study, cohort 3.
Calculate the mean radiotherapy doses to the organs at risk (salivary gland, spinal cord and brainstem) will be calculated and recorded at baseline and compared to doses from the adaptive plan at weeks 3 and 5. | Through main study treatment period, estimated 5 years.
  To calculate the mean radiotherapy doses to the organs at risk (salivary gland, spinal cord and brainstem) will be calculated and recorded at baseline and compared to doses from the adaptive plan at weeks 3 and 5 in the main study, cohort 1.

CONTACTS AND LOCATIONS:
Overall Officials: Kee H. Wong, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Head and Neck Unit, Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No